CLINICAL TRIAL: NCT00430144
Title: A Phase II Study of Belotecan (CKD-602) in Recurrent or Progressive Carcinoma of Uterine Cervix
Brief Title: Belotecan (CKD-602) in Recurrent or Progressive Carcinoma of Uterine Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sokbom Kang (Other Government)
Responsible Party: Sponsor-Investigator, Sokbom Kang, director, gynecologic oncology research branch, National Cancer Center, Korea
Organization: National Cancer Center, Korea (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-214
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — belotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CKD-602 (Experimental)
  Interventions: Drug: Belotecan(CKD-602)

INTERVENTIONS:
Drug: Belotecan(CKD-602) — Belotecan was administrated at 0.5 mg/m(2)/day for 5 consecutive days every 3-week cycle
  Other Names: Camptobel

SUMMARY:
-list item one, The purpose of this study is to evaluate the overall response rate of belotecan (CKD-602) in recurrent or progressive carcinoma of uterine cervix

DETAILED DESCRIPTION:
* list item one, to evaluate toxicities of Belotecan
* list item two, to evaluate duration of primary response for responding patients
* list item three, to evaluate time to disease progression
* list item four, to evaluate progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, patients with recurrent uterine cervical carcinoma who were unsuitable candidates for curative treatment with surgery and/or radiotherapy.
* One of the following histologic types
* Squamous cell carcinoma
* Adenocarcinoma
* Adenosquamous carcinoma
* Clinically measurable disease
* Performance status of 0, 1, 2 on the ECOG criteria

Exclusion Criteria:

* Histology of neuroendocrine tumors
* Patient previously treated with topoisomerase-I inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
overall response rate of belotecan (CKD-602) | 1 week before the start of Cycle 4, 3 weeks later Cycle 6 or at discontinuation of study treatment, and then at least every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sokbom Kang, Principal Investigator — National cancer cencer
Locations (1):
- National cancer center, Seoul, South Korea

REFERENCES:
- [Derived] Hwang JH, Lim MC, Seo SS, Park SY, Kang S. Phase II study of belotecan (CKD 602) as a single agent in patients with recurrent or progressive carcinoma of uterine cervix. Jpn J Clin Oncol. 2011 May;41(5):624-9. doi: 10.1093/jjco/hyr017. Epub 2011 Feb 24. PMID 21355002